CLINICAL TRIAL: NCT03785691
Title: Validating the Effect of Ondansetron and Mirtazapine in Treating Hyperemesis Gravidarum: A Double-Blind Randomised Placebo-Controlled Multicentre Trial
Brief Title: Validating the Effect og Ondansetron and Mirtazapine in Treating Hyperemesis Gravidarum
Acronym: VOMIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruiting difficulties
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Bispebjerg Hospital (Other); Aarhus University Hospital (Other); Herlev and Gentofte Hospital (Other); Hvidovre University Hospital (Other); Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Regionernes Medicinpulje (Unknown); Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Anne Ostenfeld, MD, PhD student, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VOMIT
Record Dates: First submitted 2018-11-13; First posted 2018-12-24 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Hyperemesis Gravidarum; Nausea Gravidarum; Vomiting of Pregnancy
Keywords: Hyperemesis Gravidarum (HG); Mirtazapine; Ondansetron; Pregnancy; Nausea and Vomiting of Pregnancy (NVP); Randomized Controlled Trial (RCT)
MeSH Terms: conditions — Hyperemesis Gravidarum; Nausea | interventions — Mirtazapine; Ondansetron

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled multicenter trial testing already marketed drugs on a new indication.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All oral tablets will be encapsulated in gelatine to ensure identical look, smell and taste.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mirtazapine (Experimental): Mirtazapine 15 mg oral tablet (incapsulated in gelatine to provide blinding) will be administered once daily (bedtime) for 7 days. Placebo (empty gelatine capsule) will be administered once daily (morning).
  On Day 7 dosage increase is optional. If desired, mirtazapine 30 mg oral tablet (incapsulated in gelatine) will be administered once daily (bedtime) for 7 days. Placebo (empty gelatine capsule) will be administered three times daily (morning, noon and late afternoon). In case dosage increase is not desired, the subject will continue the initial treatment for an additional 7 days.
  Interventions: Drug: Mirtazapine
- Ondansetron (Experimental): Ondansetron 8 mg oral tablet (incapsulated in gelatine) will be administered twice daily (morning and bedtime) for 7 days.
  On Day 7 dosage increase is optional. If desired, ondansetron 8 mg oral tablet (incapsulated in gelatine) will be administered four times daily (morning, noon, late afternoon and bedtime) for 7 days. In case dosage increase is not desired, the subject will continue the initial treatment for an additional 7 days.
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): Placebo oral tablet (empty gelatine capsule) will be administered twice daily (morning and bedtime) for 7 days.
  On Day 7 dosage increase is optional. If desired, placebo oral tablet (empty gelatine capsule) will be administered four times daily (morning, noon, late afternoon and bedtime) for 7 days. In case dosage increase is not desired, the subject will continue the initial treatment for an additional 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine 15 mg oral tablet (incapsulated in gelatine to provide blinding) will be administered once daily (bedtime) for 7 days. Placebo (empty gelatine capsule) will be administered once daily (morning).
  On Day 7 dosage increase is optional. If desired, mirtazapine 30 mg oral tablet (incapsulated in gelatine) will be administered once daily (bedtime) for 7 days. Placebo (empty gelatine capsule) will be administered three times daily (morning, noon and late afternoon). In case dosage increase is not desired, the subject will continue the initial treatment for an additional 7 days.
  Other Names: KRKA Mirtazapine Oral Tablet
  Arms: Mirtazapine
Drug: Ondansetron — Ondansetron 8 mg oral tablet (incapsulated in gelatine) will be administered twice daily (morning and bedtime) for 7 days.
  On Day 7 dosage increase is optional. If desired, ondansetron 8 mg oral tablet (incapsulated in gelatine) will be administered four times daily (morning, noon, late afternoon and bedtime) for 7 days. In case dosage increase is not desired, the subject will continue the initial treatment for an additional 7 days.
  Other Names: Bluefish Ondansetron Oral Tablet
  Arms: Ondansetron
Drug: Placebo — Placebo oral tablet (empty gelatine capsule) will be administered twice daily (morning and bedtime) for 7 days.
  On Day 7 dosage increase is optional. If desired, placebo oral tablet (empty gelatine capsule) will be administered four times daily (morning, noon, late afternoon and bedtime) for 7 days. In case dosage increase is not desired, the subject will continue the initial treatment for an additional 7 days.
  Other Names: Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
The aim is to investigate the efficacy of mirtazapine and ondansetron as treatment for hyperemesis gravidarum(HG).

The setup is a double-blind multicenter trial where patients suffering from HG will be randomized to treatment with either mirtazapine, ondansetron or placebo (1:1:1).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any trial related procedures are performed
* Female age >18 years
* Pregnant woman with gestational age between 5+0 and 19+6
* Nausea and vomiting without other obvious reason
* PUQE-24 score ≥13 OR PUQE-24 score ≥7 AND

  1. weight loss >5% of pre-pregnancy weight and/or
  2. hospitalisation due to nausea and vomiting of pregnancy
* Singleton pregnancy
* The subject must be willing and able to comply with trial protocol

Exclusion Criteria:

* Mola pregnancy, multiple gestation or non-vital pregnancy
* Nausea and vomiting of other aetiology than NVP
* Allergic to selective 5-HT3-receptor antagonists
* Ongoing treatment with antidepressant medication
* Pre-existing diagnosis of chronic kidney disease, diabetes type 1 or 2, significant cardiac disease (incl. long QT syndrome), epilepsy, HIV. In case of other pre-existing conditions subjects might be excluded based on individual assessment by an MD
* Elevated liver enzymes (ALAT>150 U/l)
* Elevated creatinine (>100 µmol/l)
* ECG showing long QT-syndrome (QTc >460msek)
* Weekly alcohol intake >2 units of alcohol
* Not able to take medicine orally
* Not able to understand spoken and/or written Danish
* Participation in another investigational drug trial within current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in nausea and vomiting from baseline to Day 2 (short term) in the mirtazapine group versus the placebo group. | 2 days
  Change in Pregnancy Unique Quantification of Emesis 24 score (PUQE-24 score) (patient reported) from baseline to Day 2 (short term) in the mirtazapine group versus the placebo group. PUQE-24 score ranges 3-15 with 3 being better and 15 being worse.
Change in nausea and vomiting from baseline to Day 2 (short term) in the ondansetron group versus the placebo group. | 2 days
  Change in PUQE-24 score (patient reported) from baseline to Day 2 (short term) in the ondansetron group versus the placebo group.
Change in nausea and vomiting from baseline to Day 14(+/-1) (long term) in the mirtazapine group versus the placebo group. | 14 days
  Change in PUQE-24 score (patient reported) from baseline to Day 14(+/-) (long term) in the mirtazapine group versus the placebo group. Only tested if outcome 1 is significant.
Change in nausea and vomiting from baseline to Day 14(+/-1) (long term) in the ondansetron group versus the placebo group. | 14 days
  Change in PUQE-24 score (patient reported) from baseline to Day 14(+/-) (long term) in the ondansetron group versus the placebo group. Only tested if outcome 2 is significant.
Change in nausea and vomiting from baseline to Day 2 (short term) in the mirtazapine group versus the ondansetron group. | 2 days
  Change in PUQE-24 score (patient reported) from baseline to Day 2 (short term) in the mirtazapine group versus the ondansetron group. Only tested if outcome 1 is significant.

SECONDARY OUTCOMES:
Change in nausea and vomiting from baseline to Day 14(+/-1) in the mirtazapine group versus the ondansetron group. | 14 days
  Change in PUQE-24 score (patient reported) from baseline to Day 14(+/-1) in the mirtazapine group versus the ondansetron group.
Overall nausea and vomiting during the intervention in the three different groups. | 14 days
  Area under the curve for PUQE-24 score (patient reported) during the intervention in the three different groups.
Change in well-being during the intervention in the three different groups. | 14 days
  Change in PUQE well-being score (patient reported) during the intervention in the three different groups.
Change in nausea during the intervention in the three different groups. | 14 days
  Change in daily nausea visual analog scale (VAS) (patient reported) during the intervention in the three different groups. VAS score ranges 0-100 with 0 being better and 100 being worse. Numbers are not visible to subjects.
Change in vomiting during the intervention in the three different groups. | 14 days
  Change in number of daily vomiting episodes (patient reported) during the intervention in the three different groups.
Occurrence of side effects in the three different groups. | 19 days
  Occurrence of side effects (patient reported and registered by trial personnel) during and until 5 days after the intervention in the three different groups.
Change in quality of life for nausea and vomiting during pregnancy from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups. | 14 days
  Change in Health-Related Quality of Life for Nausea and Vomiting during Pregnancy (NVPQOL) score (patient reported) from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups. NVPQOL score ranges 30-210 with 30 being better and 210 being worse.
Change in severity of hyperemesis gravidarum from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups. | 14 days
  Change in HyperEmesis Level Prediction (HELP) score (patient reported) from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups. HELP score ranges 0-50 with 0 being better and 50 being worse.
Change in health-related quality of life from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups. | 14 days
  Change in health status (EQ-5D-5L) (patient reported) from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups.
Change in sleep quality from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups. | 14 days
  Change in modified Pittsburg Sleep Quality Index (PSQI) (patient reported) from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups.Modified PSQI score ranges 0-12 with 0 being better and 12 being worse.
Patient satisfaction with treatment Day 7(+/-1) and Day 14(+/-1) in the three different groups. | 14 days
  Patient satisfaction with treatment VAS (patient reported) on Day 7(+/-1) and Day 14(+/-1) in the three different groups. VAS score ranges 0-100 with 0 being better and 100 being worse. Numbers are not visible to subjects.
Change in patient consideration of termination of pregnancy from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups. | 14 days
  Change in patient consideration of termination of pregnancy (patient reported) from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups.
Request for dosage increase in the three different groups. | 14 days
  Frequency of request for dosage increase in the three different groups.
Request for continuation of trial medication after end of intervention in the three different groups. | 14 days
  Frequency of request for continuation of trial medication after end of intervention in the three different groups.
Use of rescue medication during the intervention in the three different groups. | 14 days
  Use of rescue medication during (patient reported) the intervention in the three different groups.
Number of days on sick leave during the intervention in the three different groups | 14 days
  Number of days on sick leave (patient reported) during the intervention in the three different groups
Necessity of i.v.-fluids during the intervention in the three different groups. | 14 days
  Amount of treatments with i.v.-fluids during the intervention in the three different groups.
Need of hospitalisation during the intervention in the three different groups. | 14 days
  Number of days of hospitalisations during the intervention in the three different groups.
Weight change from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups. | 14 days
  Weight change in kg from baseline to Day 7(+/-1) and baseline to Day 14(+/-1) in the three different groups.
Pregnancy outcome: Live birth, loss or termination of pregnancy | 8 months
  Live birth, loss or termination of pregnancy.
Delivery outcome: Mode of delivery | 8 months
  Mode of delivery: Vaginal, cesarian, vacuum extraction.
Delivery outcome: Delivery complications | 8 months
  Eg. postpartum hemorrhage, shoulder dystocia, sphincter rupture
Live birth outcome: birth weight. | 8 months
  Birth weight in g.
Live birth outcome: gestational age at birth. | 8 months
  Gestational age at birth in weeks plus days.
Live birth outcome: APGAR score. | 8 months
  APGAR score at 1, 5 and 10 minutes after birth. APGAR score ranges 0-10 with 0 being worse and 10 being better.
Live birth outcome: umbilical cord pH. | 8 months
  Umbilical cord pH at birth.
Live birth outcome: placenta weight. | 8 months
  placenta weight in g.
Live birth outcome: sex. | 8 months
  offsprings sex.
Live birth outcome: hospitalizations on neonatal ward during the first month post-partum. | 9 months
  Hospitalizations of the offspring in neonatal ward during the first month post-partum.
Live birth outcome: congenital malformations (depending on gestational age also registered on early ended pregnancies). | 8 months
  Congenital malformations.
Occurrence of treatment failure in the three different groups. | 14 days
  Frequency of and time to treatment failure in the three different groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Ostenfeld, MD, Principal Investigator — Department of Obstetrics and gynecology, Nordsjællands Hospital Hillerød
Locations (7):
- Denmark (7):
  - Department of Gynaecology and Obstetrics, Aarhus University Hospital, Aarhus
  - Department of Gynaecology and Obstetrics, Rigshospitalet, Copenhagen
  - Department of Gynaecology and Obstetrics, Herlev Hospital, Herlev
  - Department of Gynaecology and Obstetrics, Nordsjællands Hospital, Hillerød
  - Department of Gynaecology and Obstetrics, Hvidovre Hospital, Hvidovre
  - Department of Gynaecology and Obstetrics, Kolding Sygehus, Kolding
  - Department of Gynaecology and Obstetrics, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
Access to patient level data and supporting clinical documents may be requested. Requests will be reviewed on the basis of methodological proposal. Patient data will be de-identified to protect the privacy of trial patients in line with applicable laws and regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication, no end date.

REFERENCES:
- [Derived] Ostenfeld A, Carlsen SE, Jensen AK, Futtrup TB, Westergaard HB, Pedersen LH, Andersen JT, Petersen TS, Lokkegaard ECL; VOMIT investigation group. Mirtazapine or ondansetron for hyperemesis gravidarum: a randomized placebo-controlled trial. Am J Obstet Gynecol. 2025 Dec 30:S0002-9378(25)00982-2. doi: 10.1016/j.ajog.2025.12.061. Online ahead of print. PMID 41478546
- [Derived] Ostenfeld A, Petersen TS, Futtrup TB, Andersen JT, Jensen AK, Westergaard HB, Pedersen LH, Lokkegaard ECL. Validating the effect of Ondansetron and Mirtazapine In Treating hyperemesis gravidarum (VOMIT): protocol for a randomised placebo-controlled trial. BMJ Open. 2020 Mar 24;10(3):e034712. doi: 10.1136/bmjopen-2019-034712. PMID 32209630

DOCUMENTS (4):
  • Study Protocol: Current version (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT03785691/Prot_000.pdf
  • Study Protocol: Original version (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT03785691/Prot_001.pdf
  • Statistical Analysis Plan: Current version (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT03785691/SAP_002.pdf
  • Statistical Analysis Plan: Original version (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT03785691/SAP_003.pdf